CLINICAL TRIAL: NCT05205005
Title: Targeting the Endothelial Glycocalyx to Enhance Vascular Function and Exercise-Induced Vascular Adaptations in Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CARB-005-21S
Record Dates: First submitted 2021-12-20; First posted 2022-01-24 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Endothelial function; Glycocalyx; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Dietary supplement vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary supplementation of glycocalyx precursors (DSGP) (Experimental): Participants will daily ingest 3,712mg (i.e., six capsules) of DSGP for eight weeks. DSGP, commercially available as Endocalyx (Microvascular Health Solutions LLC, Alpine, UT), include glucosamine sulfate, fucoidan, superoxide dismutase, and high molecular weight hyaluronan.
  Interventions: Drug: Endocalyx
- Placebo (Placebo Comparator): Participants will daily ingest 6 capsules daily of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Endocalyx — 3,712mg (six capsules) of DSGP for eight weeks.
  Arms: Dietary supplementation of glycocalyx precursors (DSGP)
Drug: Placebo — Ingredients per capsule (6 capsules per day) Nu-Mag Nat 10.00mg Rice Flour White 830 mg Magnesium Stearate 10.00mg
  Arms: Placebo

SUMMARY:
The prevalence of type 2 diabetes (T2D) continues to increase in the US, with 26.8 million adults carrying a diagnosis. Importantly, T2D is widespread in the Veteran population. This epidemic of T2D also contributes to the staggering rates of cardiovascular disease and cardiovascular mortality. Lifestyle modifications, including increased physical activity, are recommended as first-line therapy for the management of T2D. Unfortunately, patients with T2D exhibit diminished vascular adaptations to exercise. The proposed project will test the overall hypothesis that degradation of the endothelial glycocalyx, a characteristic feature of T2D, precludes shear stress mechanotransduction and consequent exercise-induced vascular adaptations. As such, the investigators pose that restoration of the endothelial glycocalyx via dietary supplementation of glycocalyx precursors will potentiate vascular adaptations to exercise in Veterans with T2D.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2D) continues to increase in the US. Importantly, T2D is widespread among Veterans. This T2D epidemic also contributes to the staggering rates of cardiovascular disease (CVD) and cardiovascular mortality. Current standards of medical care for T2D emphasize prioritizing the use of therapies that decrease CVD risk. Lifestyle modifications, such as increased physical activity, are recommended as first-line therapy for the management of T2D. Unfortunately, the efficacy of these interventions for preventing CVD morbidity and mortality in patients with T2D remains questionable. Evidence indicates that exercise training in T2D subjects does not elicit optimal vascular adaptations, including improvements in endothelial function. It is likely that such lessened vascular adaptations explain why increased physical activity does not lead to a robust reduction in CVD morbidity and mortality in T2D. A better understanding of the mechanisms responsible for the deficit of vascular adaptations to exercise in T2D is required for identifying new adjuvant therapeutics aimed at maximizing the cardiovascular benefits of exercise.

The primary goal of this project is to establish the endothelial glycocalyx as a novel target organ for heightening exercise-induced vascular adaptations. To that end, a dietary supplement that contains glycocalyx precursors (glucosamine sulfate, fucoidan, superoxide dismutase, and high molecular weight hyaluronan) will be used as an innovative "tool" to restore the endothelial glycocalyx in T2D subjects. Demonstration that dietary supplementation of glycocalyx precursors (DSGP) is effective at enhancing endothelial glycocalyx integrity in patients with T2D will be accomplished in the Proof of Concept Clinical Trial Phase (or Aim 1) of this project. Subsequently, in the Expended Clinical Trial Phase (or Aim 2), the use of the DSGP will allow us to test the hypothesis that glycocalyx restoration re-sensitizes the endothelium to shear stress mechanotransduction and thus potentiates exercise-induced vascular adaptations. This project will be the first to determine if targeting the glycocalyx is a viable therapeutic strategy for boosting exercise-induced endothelial benefits in diabetes.

The overarching hypothesis is that endothelial glycocalyx degradation is a key factor that precludes shear stress mechanotransduction and consequent exercise-induced vascular adaptations in T2D. A corollary to this hypothesis is that restoration of the endothelial glycocalyx by DSGP will improve vascular adaptations to exercise in T2D.

Specific aims are as follows:

Aim 1 (Proof of Concept Clinical Trial Phase): Document that DSGP enhances endothelial glycocalyx integrity in Veterans with T2D. The effects of DSGP for eight weeks on glycocalyx integrity and endothelial function will be studied using a double-blinded randomized placebo control trial. Sample size = 24 subjects (12 per group) for Aim 1.

Aim 2 (Expanded Clinical Trial Phase): Demonstrate the permissive role of the endothelial glycocalyx for exercise-induced vascular adaptations in Veterans with T2D. Having shown that endothelial glycocalyx restoration via DSGP in T2D subjects is feasible, will now investigate whether such supplementation potentiates exercise training-induced improvements in endothelial function. This will be accomplished with a factorial balanced design in which T2D subjects will be randomized to DSGP or placebo with and without concurrent exercise training for eight weeks. Sample size = 72 subjects (18 per group).

ELIGIBILITY:
Inclusion Criteria:

1. 45-74 years of age at the time of enrollment
2. Diagnosis of T2D by a health care provider, confirmed by chart review
3. HbA1c <9% and fasting blood glucose <200 mg/dL at screening visit
4. Body mass index (BMI) 25-45 kg/m2
5. Women should be postmenopausal (absence of menses for at least 1 year)
6. Sedentary subjects (<2 days/week of vigorous exercise)
7. Willingness to follow up instructions provided by study team

Exclusion Criteria:

Exclusion:

1. Evidence of cardiac arrhythmias, unstable angina (or other cardiac event), heart failure or stroke in the last 12 months
2. Evidence of chronic kidney disease stage IV or V (GFR <30 mL/min)
3. Evidence of uncontrolled hypertension, systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg on more than 2 occasions in the past 12 months or at screening visit
4. Diagnosis of chronic liver disease
5. Uncontrolled thyroid dysfunction (abnormal TSH within 3 months of study enrollment)
6. Active cancer
7. Current use of hormone replacement therapy
8. Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
9. Current pregnancy or intent to become pregnant during the course of the study
10. Inability to swallow capsules
11. Known allergies to any of the compounds in the supplement: glucosamine extract, fucoidan extract, olive extract, artichoke extract, red and white grapes extract, melon concentrate, hyaluronic acid

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camila Margarita M Manrique Acevedo, MD, Principal Investigator — Harry S. Truman Memorial, Columbia, MO
Locations (1):
- Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Details of research products in this project will be in text, table, plots and images that will be disseminated in peer reviewed journals and/or conference proceedings. Datasets that underlie these research products will be made available upon reasonable written request and review with the ACOS/R&D and the ISSO within a reasonable time
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon completion of data analysis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This clinical trial is a proof of concept clinical trial phase that corresponds to Aim 1 of a larger project. The participants assigned to intervention in this trial completed either the DSGP supplementation or placebo arms. No aim 2/clinical trial phase 2 will be enacted for the larger project.
Groups:
- Placebo: Participants will daily ingest 6 capsules daily of placebo for eight weeks.
  Placebo: Ingredients per capsule (6 capsules per day) Nu-Mag Nat 10.00mg Rice Flour White 830 mg Magnesium Stearate 10.00mg
Period: Overall Study
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 9 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.0) | 60.6 (8.4) | 63.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Glygocalyx Integrity - Perfused Boundary Region
Description: Glycocalyx integrity will be assessed non-invasively using the GlycoCheck. The Glycocheck video microscope instrument will be placed under the subject's tongue to assess red blood cell penetration of the glycocalyx lining. PBR (perfused boundary region) is a measure of distance (mcm) that red blood cells penetrate into the glycocalyx. An increase in PBR in indicative of lower glycocalyx integrity.
Time Frame: Change from baseline to eight weeks assessment
Population: participants that completed full study intervention with baseline and eight week assessment.
Measure: Mean (Standard Error); unit: Delta micrometers (mcm)
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
Number analyzed (Participants) | 10 | 12
Delta micrometers (mcm) | 0.11 (0.17) | -0.16 (0.15)

2. Secondary Outcome: Brachial Artery Flow Mediated Dilation
Description: Arterial measurements will be performed by imaging the brachial artery artery longitudinally using high-resolution duplex ultrasonography. Arterial vasodilatory responses to hyperemia (flow-mediated dilation; FMD) will be examined by inflating a cuff up to 250 mmHg for five minutes. Before, during and after rapid release of the cuff, brachial artery blood flow velocity and diameter will be continuously measured. This is a measurement of endothelial function. When assessing FMD, the cuff will squeeze the arm tightly; however, any discomfort will be alleviated as soon as the pressure in the cuff is released.
Time Frame: Baseline and final assessment (Week 8)
Population: participants that completed full study intervention with baseline and eight week assessment.
Measure: Mean (Standard Error); unit: FMD %
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
Number analyzed (Participants) | 10 | 12
FMD %
  Baseline | 2.93 (0.39) | 2.14 (0.27)
  Final | 3.20 (0.47) | 1.87 (0.34)

3. Secondary Outcome: Insulin-stimulated Leg Blood Flow
Description: Insulin-stimulated leg blood flow will be assessed via Doppler and contrast-enhanced ultrasound during an insulin-dextrose clamp. After a minimum of 20 minutes in supine rest, baseline cardiovascular measurements will be collected, including Doppler and contrast-enhanced ultrasound-based measures, blood samples obtained and then the insulin clamp will start. Briefly, insulin (Humulin R U-100) will be infused via IV at a constant rate of 80mU/m2 body surface area/min for the three-hour period. Blood glucose will be measured at five-minute intervals and maintained at fasting levels; this will be achieved by variable IV infusion rates of a 20% dextrose solution. The measurements described will allow for the assessment of the insulin stimulated leg blood flow
Time Frame: Baseline and final assessment (Week 8)
Population: participants that completed full study intervention with baseline and eight week assessment.
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
Number analyzed (Participants) | 10 | 12
mL/min
  Baseline | 5.98 (11.92) | 16.93 (15.38)
  Final | 2.97 (12.14) | 9.55 (9.03)

4. Secondary Outcome: Femoral Artery Flow Mediated Dilation
Description: Arterial measurements will be performed by imaging the femoral artery longitudinally using high-resolution duplex ultrasonography. Arterial vasodilatory responses to hyperemia (flow-mediated dilation; FMD) will be examined by inflating a cuff up to 250 mmHg for five minutes. Before, during and after rapid release of the cuff, femoral artery blood flow velocity and diameter will be continuously measured (these are used to calculate the FMD). This is a measurement of endothelial function. When assessing FMD, the cuff will squeeze the leg tightly; however, any discomfort will be alleviated as soon as the pressure in the cuff is released.
Time Frame: Baseline and final assessment (Week 8)
Population: participants that completed full study intervention with baseline and eight week assessment.
Measure: Mean (Standard Error); unit: FMD %
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
Number analyzed (Participants) | 10 | 12
FMD %
  Baseline | 2.93 (0.39) | 2.14 (0.27)
  Final | 3.20 (0.47) | 1.87 (0.34)

ADVERSE EVENTS:
Time Frame: Screening visit until final assessment (week 8 assessment)
Arm/Group | Dietary Supplementation of Glycocalyx Precursors (DSGP) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary Supplementation of Glycocalyx Precursors (DSGP) (N=12) | Placebo (N=12)
Tendon injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant reported an Achilles tendon injury
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant reported "loose stools"
Stomach Ache (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant reported "upset stomach"
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Participant reported headache
PT/PTT lab elevation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — PT/PTT were elevated compared with baseline
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Participant reported experiencing "itchiness"
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant reported experiencing hemorrhoids

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05205005/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT05205005/ICF_002.pdf